CLINICAL TRIAL: NCT01820481
Title: Double Blinded, Randomized, Placebo Controlled, Multi-center, Phase 2 : Exploratory Clinical Study to Evaluate the Efficacy, Dose-response and Safety of WIN-901X in Asthma Patients
Brief Title: Safety and Efficacy of WIN-901X in Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Whanin Pharmaceutical Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WIN-901X-P2
Record Dates: First submitted 2013-03-25; First posted 2013-03-28 (Estimated); Last update posted 2013-12-09 (Estimated); Status verified 2013-12

CONDITIONS: Asthma
Keywords: Asthma; Bronchial Diseases; Respiratory Tract Diseases; Lung Diseases, Obstructive; Lung Diseases
MeSH Terms: conditions — Asthma; Bronchial Diseases; Respiratory Tract Diseases; Lung Diseases, Obstructive; Lung Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Treatment 1 (Experimental)
  Interventions: Drug: WIN-901X dose level 1
- Treatment 2 (Experimental)
  Interventions: Drug: WIN-901X dose level 2
- Treatment 3 (Experimental)
  Interventions: Drug: WIN-901X dose level 3
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: WIN-901X dose level 1 — 100mg Bid, PO, 12weeks
  Arms: Treatment 1
Drug: WIN-901X dose level 2 — 200mg Bid, PO, 12weeks
  Arms: Treatment 2
Drug: WIN-901X dose level 3 — 300mg Bid, PO, 12weeks
  Arms: Treatment 3
Drug: Placebo — Bid, PO, 12weeks
  Arms: Placebo

SUMMARY:
This clinical trial is designed to evaluate the efficacy, dose-response and safety of WIN-901X in Asthma patients.

DETAILED DESCRIPTION:
Double blinded, Randomized, Placebo Controlled, Multi-center, Phase 2 : Exploratory Clinical Study to Evaluate the Efficacy, Dose-response and Safety of WIN-901X in Asthma Patients

ELIGIBILITY:
Inclusion Criteria:

* Greater than or equal to 20 and less than 80 years of age
* Have physician diagnosed asthma with irreversible airway obstruction at least 6 months prior to the screening
* FEV1 between 60% and 85% before inhaling fast-acting bronchodilator at screening
* No history of smoking at least one year prior to the screening
* Having voluntarily signed an informed consent

Exclusion Criteria:

* Have visited emergency room due to the worsening asthma symptoms, within 4 weeks before the screening
* Have been hospitalized due to an acute worsening of asthma within 3 months before the screening
* Have a history of laryngitis, pyrexia, sinusitis, otitis media, respiratory tract infection, and infectious rhinitis within 4 weeks prior to the screening
* Have malignant tumor

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 209 (Actual)
Dates: Start 2012-09; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Compare the change of FEV1% to the baseline after the medication | Baseline, week 12
  FEV1: Forced Expiratory Volume In One Second

SECONDARY OUTCOMES:
Compare the change of ACQ to the baseline after the medication | Baseline, week 12
  ACQ: Asthma Control Questionnaire
Ratio of the date, where no rescue drug was used, during the trial | Baseline, week 12
Ratio of symptom free days during the trial | Baseline, week 12

CONTACTS AND LOCATIONS:
Overall Officials: Park Hae Sim, M.D., Professor, Study Chair — Yes
Locations (1):
- Ajou University Medical Center, Suwon, South Korea